CLINICAL TRIAL: NCT01590667
Title: Double-blind, Randomized, Placebo-controlled, Crossover Clinical Investigation to Evaluate the Effect of Litramine on Fecal Fat Excretion in Healthy Subjects
Brief Title: Effect of Litramine on Fat Excretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: INQ/028711
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Subjects
Keywords: Fat excretion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Litramine (Active Comparator): 2 tablets 3 times daily (oral consumption, 30 minutes after meal)
  Interventions: Device: Litramine
- Placebo (Placebo Comparator): 2 tablets 3 times daily (oral consumption, 30 minutes after meal)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Litramine — 2 tablets 3 times daily (oral consumption, 30 minutes after meal)
  Arms: Litramine
Device: Placebo — 2 tablets 3 times daily (oral consumption, 30 minutes after meal)
  Arms: Placebo

SUMMARY:
The study aims to evaluate the effect of Litramine on fecal fat excretion in healthy subjects, to provide more comprehensive and robust clinical evidence in its mode of action for the treatment of obesity and weight management through dietary fat binding.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-30 kg/m2
* Accustomed to 3 main meals/day
* Commitment to avoid the use of other weight management products during study
* Females' agreement to use appropriate birth control methods during the active study period
* Self-reported regular bowel movement (1-2 times per day)
* Subject declares in writing his/her consent to participate, understands requirements of the study and is willing to comply

Exclusion Criteria:

* Known sensitivity to the ingredients of the device
* Diabetes mellitus (type 1 or 2)
* History or clinical signs of endocrine disorders
* Clinically relevant excursions of safety parameter
* Current use of anti-depressants
* Presence of acute or chronic gastrointestinal disease
* Uncontrolled hypertension (more than 160/110 mm Hg)
* Stenosis in the gastrointestinal tract
* Bariatric surgery
* Abdominal surgery within the last 6 months prior to enrollment
* History of eating disorders such as bulimia, anorexia nervosa within the past 12 months
* Other serious organ or systemic diseases such as cancer
* Any medication that could influence gastrointestinal functions
* Pregnancy or nursing
* Any medication or use of products for the treatment of obesity within 6 weeks prior to enrolment
* History of abuse of drugs, alcohol or medication
* Presence of other factor(s) that, in the investigator's judgment, should preclude subject participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Difference between Litramine and placebo in changes of percentage fecal fat excretion after intervention | 7 days per intervention
  The amount of fat excreted in the feces will be quantified by the near-infrared reflectance analysis (NIRA)

SECONDARY OUTCOMES:
Full blood count | Approximately 45 days
  Analysis of hemoglobin, hematocrit, erythrocytes, thrombocytes, and leucocytes
Clinical chemistry | Approximately 45 days
  Liver function, renal function, protein metabolism, lipid metabolism
Blood pressure | Approximately 45 days
  Sitting blood pressure and heart rate will be measured using standard devices

CONTACTS AND LOCATIONS:
Overall Officials: Regina Busch, MD, Principal Investigator — analyze & realize AG
Locations (1):
- Weißenseer Weg 111, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Uebelhack R, Busch R, Alt F, Beah ZM, Chong PW. Effects of cactus fiber on the excretion of dietary fat in healthy subjects: a double blind, randomized, placebo-controlled, crossover clinical investigation. Curr Ther Res Clin Exp. 2014 Jun 21;76:39-44. doi: 10.1016/j.curtheres.2014.02.001. eCollection 2014 Dec. PMID 25067985